CLINICAL TRIAL: NCT00002159
Title: A Randomized, Open, Comparative Multicenter Study of Initial Treatment With Intravenous Itraconazole Versus Amphotericin B Followed by Consolidation Treatment With Itraconazole Capsules in Patients With Blastomycosis or Histoplasmosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 254A; ITR-USA-118
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-12

CONDITIONS: HIV Infections; Histoplasmosis; Blastomycosis
Keywords: Itraconazole; Histoplasmosis; Antifungal Agents; Acquired Immunodeficiency Syndrome; Amphotericin B; AIDS-Related Complex; Blastomycosis; Antibiotics, Antifungal
MeSH Terms: conditions — HIV Infections; Histoplasmosis; Blastomycosis; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Itraconazole; Amphotericin B

INTERVENTIONS:
Drug: Itraconazole
Drug: Amphotericin B

SUMMARY:
To assess the safety of intravenous itraconazole compared to amphotericin B in HIV positive or negative persons with blastomycosis or histoplasmosis.

DETAILED DESCRIPTION:
Patients are randomized to receive IV itraconazole for 2 days, then either itraconazole daily for 5 days or amphotericin B daily for 7 days. IV treatment is followed by consolidation with oral itraconazole for up to 1 year.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positive or negative status.
* Blastomycosis or histoplasmosis.
* Life expectancy of at least 1 week.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Liver disease.
* Self-limiting fungal disease.
* Very severe fungal disease such as meningeal involvement.
* Acute respiratory disease.

Concurrent Medication:

Excluded at any time:

* Terfenadine.
* Astemizole.
* Oral midazolam.
* Triazolam.
* Cisapride.
* Phenytoin.
* Phenobarbital.
* Rifampin.
* Rifabutin.

Excluded during oral consolidation:

* H2 blockers.
* Chronic antacids.
* Omeprazole.
* Lansoprazole.

Patients with the following prior condition are excluded:

Hypersensitivity to azole antifungals.

Prior Medication:

Excluded at any time:

More than 3 days of amphotericin B, fluconazole, or ketoconazole.

Excluded within 2 weeks prior to study entry:

* Phenytoin.
* Phenobarbital.
* Rifampin.
* Rifabutin.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UAB Station / Infectious Division, Birmingham, Alabama
  - Univ of Arkansas for Med Sciences, Little Rock, Arkansas
  - Division of Infectious Diseases, Atlanta, Georgia
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Community Hosp, Indianapolis, Indiana
  - LSU Med Ctr / Div of Pulmonary & Critical Care Med, Shreveport, Louisiana
  - Ann Arbor Veterans Administration Med Ctr, Ann Arbor, Michigan
  - Univ of Missouri / Division of Infectious Diseases, Kansas City, Missouri
  - Infectious Diseases Association / Research Med Ctr, Kansas City, Missouri